CLINICAL TRIAL: NCT03343379
Title: Core Stability as a Risk Factor for the Development of Lower Extremity Injuries: a Prospective Study
Brief Title: Core Stability Measures as a Risk Factor for the Development of Lower Extremity Injuries in Physical Education Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014/0780
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Leg Injuries
Keywords: Abdominal muscles; Back muscles; Core stability; Field test; Muscle strength dynamometer; Lower extremity injury; Risk assessment; Prospective studies
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Intervention Model Description: 1 group of participants was screened at the start of the study and followed prospectively for 2 years
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy cohort (Other): Core stability test
  Interventions: Other: Core stability tests

INTERVENTIONS:
Other: Core stability tests — A test battery comprised of field tests to evaluate core stability

SUMMARY:
Male and female physical education students were subjected to a clinical test battery comprised of valid and reliable tests to measure different aspects of core stability at the start of the study. After a period of 2 months testing, the injury registration procedure started with the use of an online injury registration platform and regular call back moments. After 2 years of injury registration, all data was gathered and will be analysed statistically to link the measured core stability aspects as risk factors for certain lower extremity injuries.

DETAILED DESCRIPTION:
September 2014 - December 2014: 139 male and female participants 18+ were subjected to different test to evaluate corresponding aspects of core stability. The following test were performed: Star excursion balance test; Lumbopelvic proprioception test; Lumbopelvic neuromuscular control test; Lateral step down test; Hip strength test measured with a handheld dynamometer(flexion/extension/abduction/adduction/internal rotation/external rotation); Trunk strength tests measured with a handheld dynamometer (trunk flexion and trunk extension) and core muscle endurance tests (prone bridging test/Biering-Sorenson test/side bridging tests).

January 2015 - April 2017: Prospective follow up of lower extremity injury contracted during sports activity. The injuries were confirmed by a medical examiner and were recorded in an online injury registry platform (Survey Monkey).

Statistical analysis will be performed to evaluate which core stability outcome measure can be considered a risk factor for the development of lower extremity injuries.

ELIGIBILITY:
Inclusion Criteria:

- 1st year of physical education study (enrolled at the Artevelde graduate school or the Ghent graduate school

Exclusion Criteria:

* Musculoskeletal injury at the time of study participation
* Pre-existing lower back injury
* Pre-existing lower extremity injury (less than 6 months prior to study participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Core muscle strength | 2 hours
  Isometric strength of trunk flexor and trunk extensor musculature measured in Newton
Hip strength | 2 hours
  Isometric strength of hip flexor, hip extensor, hip abductor, hip adductor and hip rotator muscles measured in Newton
Postural control | 2 hours
  Anterior, posterolateral and posteromedial reaching distance during unipodal stance, measured in cm
Core muscle endurance | 2 hours
  Endurance capacity of ventral, dorsal and lateral core musculature, measured in seconds
Sensorimotor control of core musculature | 2 hours
  Propriocention and neuromuscular control of the lumbopelvic muscles using a qualitative assessment sheet

SECONDARY OUTCOMES:
Injury history | 2 hours
  Previous lower extremity injuries, recorded using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roosen, PT, PhD, Principal Investigator — University Ghent
Locations (1):
- Vakgroep REVAKI (Ghent University - Ghent University hospital), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared after completion of the study

REFERENCES:
- [Background] De Blaiser C, De Ridder R, Willems T, Danneels L, Vanden Bossche L, Palmans T, Roosen P. Evaluating abdominal core muscle fatigue: Assessment of the validity and reliability of the prone bridging test. Scand J Med Sci Sports. 2018 Feb;28(2):391-399. doi: 10.1111/sms.12919. Epub 2017 Jun 28. PMID 28544083
- [Background] De Blaiser C, Roosen P, Willems T, Danneels L, Bossche LV, De Ridder R. Is core stability a risk factor for lower extremity injuries in an athletic population? A systematic review. Phys Ther Sport. 2018 Mar;30:48-56. doi: 10.1016/j.ptsp.2017.08.076. Epub 2017 Aug 24. PMID 29246794
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Willson JD, Dougherty CP, Ireland ML, Davis IM. Core stability and its relationship to lower extremity function and injury. J Am Acad Orthop Surg. 2005 Sep;13(5):316-25. doi: 10.5435/00124635-200509000-00005. PMID 16148357